CLINICAL TRIAL: NCT07027332
Title: Assesment of Liver Functions in Women With Polycystic Ovary Syndrome Using Fibroscan
Brief Title: Liver Stiffness And Steatosis Assessment In Women With Polycystic Ovary Syndrome Using Fibroscan
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: E-54022451-050.04-153866
Record Dates: First submitted 2025-05-28; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Polycystic Ovary Syndrome; Non-Alcoholic Fatty Liver Disease
Keywords: fibroscan; infertility; Polycystic Ovary Syndrome; Hepatic Steatosis
MeSH Terms: conditions — Polycystic Ovary Syndrome; Non-alcoholic Fatty Liver Disease; Infertility; Fatty Liver

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- PCOS Group: Women aged 18 to 45 diagnosed with Polycystic Ovary Syndrome (PCOS) according to Rotterdam criteria. Participants presented with symptoms such as menstrual irregularities, acne, or hirsutism. Exclusion criteria included alcohol consumption >20 g/day, liver disease history, pregnancy, lactation, and medication affecting liver/metabolism. Evaluations included anthropometric measurements (BMI, waist and hip circumference, waist-to-hip ratio), laboratory analyses (fasting glucose, insulin, lipid profile, liver enzymes, bilirubin fractions), hormonal assays (FSH, LH, AMH, estradiol, total and free testosterone, SHBG), ovarian ultrasonography (transabdominal or transvaginal), and liver assessment via FibroScan elastography. No interventions were administered as this was an observational study.
  Interventions: Diagnostic Test: FibroScan® (Echosens, Paris, France)
- Control Group ( Healthy, NON PCOS): Age and BMI matched healthy women aged 18 to 45 with regular menstruation for at least two years, no clinical signs of hyperandrogenism, and no history of endocrine, hepatic, renal, cardiovascular, or oncologic diseases. Participants underwent the same evaluations as the PCOS group, including anthropometric measurements, laboratory and hormonal assays, ovarian ultrasonography, and FibroScan liver elastography. No interventions were administered.
  Interventions: Diagnostic Test: FibroScan® (Echosens, Paris, France)

INTERVENTIONS:
Diagnostic Test: FibroScan® (Echosens, Paris, France) — A non-invasive liver elastography device used for clinical assessment. Liver steatosis and stiffness are measured in participants using the FibroScan device.

SUMMARY:
Polycystic Ovary Syndrome (PCOS) is a complex endocrine and metabolic disorder prevalent among women of reproductive age. It is closely associated with insulin resistance, obesity, and metabolic dysfunction, often leading to hepatic steatosis (fatty liver). This single-center, cross-sectional, case-control study evaluates liver function in PCOS patients using FibroScan, a non-invasive elastography technique. Eighteen women diagnosed with PCOS according to Rotterdam criteria and 18 age- and BMI-matched healthy controls aged 18-45 years were included. The study aims to determine whether PCOS independently affects hepatic steatosis and to assess the clinical applicability of FibroScan in this population. The results may inform early metabolic risk detection and improve multidisciplinary management strategies for PCOS.

DETAILED DESCRIPTION:
This prospective, cross-sectional study was conducted at Bezmialem Vakif University Hospital. The study included 36 women between the ages of 18 and 45. Eighteen participants were diagnosed with Polycystic Ovary Syndrome (PCOS) according to the Rotterdam 2003 criteria, which require at least two of the following features: oligo- or anovulation, clinical or biochemical hyperandrogenism, or polycystic ovarian morphology, with other endocrine disorders excluded. The remaining 18 participants, matched for age and body mass index (BMI), constituted the healthy control group.

All evaluations were conducted according to a standardized protocol approved by the university ethics committee. Each participant underwent physical examination and anthropometric assessment, including measurement of height, weight, waist and hip circumferences, and calculation of BMI and waist-to-hip ratio. Clinical hyperandrogenism was assessed using the modified Ferriman-Gallwey score by an experienced gynecologist. Participants were also evaluated for acne and androgenic alopecia. Pelvic ultrasonography was performed transabdominally or transvaginally between days 2 and 5 of the menstrual cycle, depending on anatomical and personal factors. Ovarian volume was calculated using the ellipsoid formula, and participants with structural abnormalities or dominant follicles larger than 10 mm were excluded.

Fasting venous blood samples were collected after a 13-hour overnight fast. Biochemical tests included fasting glucose, insulin, lipid profile (total cholesterol, LDL-C, HDL-C, triglycerides), liver function tests including AST (aspartate aminotransferase), ALT (alanine aminotransferase), ALP (alkaline phosphatase), GGT (gamma-glutamyl transferase), and bilirubin fractions. Renal function markers included creatinine, blood urea nitrogen, and estimated glomerular filtration rate. Additional measurements included albumin, uric acid, and platelet count. Thyroid function was assessed with thyroid-stimulating hormone (TSH), free triiodothyronine (free T3), and free thyroxine (free T4). Hormonal assays, performed between days 3 and 5 of the menstrual cycle, included follicle-stimulating hormone (FSH), luteinizing hormone (LH), estradiol (E2), anti-Müllerian hormone (AMH), total and free testosterone, sex hormone-binding globulin (SHBG), prolactin, and the free androgen index. Insulin resistance was calculated using the HOMA-IR formula.

Liver steatosis and stiffness were measured using Vibration-Controlled Transient Elastography (FibroScan®, Echosens, Paris) following at least 12 hours of fasting. All procedures were performed by a senior hepatologist blinded to the clinical and laboratory findings. CAP (Controlled Attenuation Parameter) values were used to evaluate hepatic fat content, and liver stiffness was measured in kilopascals (kPa). Measurements followed strict quality control standards including a minimum of 10 valid acquisitions, a success rate of 60% or higher, and an interquartile-to-median ratio of 0.30 or lower. CAP and stiffness cut-off values were applied according to published clinical thresholds.

To exclude secondary hepatic or endocrine conditions, all participants were screened for viral hepatitis (HBsAg, Anti-HCV, HCV RNA), HIV (Anti-HIV ELISA), and abnormal thyroid or renal function. Individuals with a history of liver disease, viral hepatitis, hepatotoxic drug use, ALT levels greater than twice the upper limit of normal for more than three months, or a personal or first-degree family history of liver cancer or autoimmune liver disorders were excluded. Pregnant or breastfeeding women were also not included.

The aim of this study is to evaluate whether PCOS independently contributes to hepatic steatosis, beyond known factors such as obesity and insulin resistance, and to assess the clinical utility of FibroScan as a non-invasive liver assessment tool in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 18 to 45 years
* Voluntary participation and signed informed consent
* For the PCOS group: diagnosis of Polycystic Ovary Syndrome (PCOS) based on the Rotterdam 2003 criteria, including at least two of the following: (1) oligo- or anovulation, (2) clinical or biochemical hyperandrogenism, (3) polycystic ovarian morphology on ultrasound
* For the control group: regular menstrual cycles in the past two years and absence of clinical or biochemical hyperandrogenism
* No history of endocrine, metabolic, hepatic, renal, cardiovascular, or oncologic disease
* Willingness and ability to undergo blood sampling, ultrasound, and FibroScan evaluations
* Ability to comply with study procedures and availability throughout the study period

Exclusion Criteria:

* Pregnancy or lactation
* Use of hormonal contraceptives, insulin sensitizers, or hepatotoxic medications within the past 3 months
* Diagnosis of diabetes mellitus, thyroid dysfunction, Cushing's syndrome, or congenital adrenal hyperplasia
* ALT ≥2 times the upper limit of normal (ULN) or single ALT >80 U/L at screening
* Positive screening for hepatitis B surface antigen (HBsAg), hepatitis C virus RNA (HCV RNA), or HIV
* History or current diagnosis of liver disease, autoimmune hepatitis, Wilson's disease, or alpha-1 antitrypsin deficiency
* Alcohol intake exceeding 20 grams per day
* Presence of ovarian cysts, endometriomas, or adnexal masses interfering with ultrasound interpretation
* Personal or first-degree family history of liver cancer or any malignancy
* Inability to understand or sign informed consent or to adhere to study requirements

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This single-center, cross-sectional, comparative study was conducted at Bezmialem Vakif University Hospital. The study population consists of women aged 18 to 45 years diagnosed with PCOS according to Rotterdam criteria and age- and BMI-matched healthy controls without endocrine or metabolic disorders.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2024-05-29 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-03-08 (Actual)

PRIMARY OUTCOMES:
Liver Steatosis Measured by Controlled Attenuation Parameter (CAP) | At baseline (single time point during study visit)
  Non-invasive quantification of hepatic steatosis in women with PCOS and controls using FibroScan elastography.

SECONDARY OUTCOMES:
Liver Stiffness Measurement (E) | At baseline (single time point during study visit)
  Assessment of liver fibrosis via liver stiffness measurement using FibroScan in PCOS and control groups.
Insulin Resistance Index (HOMA-IR) | At baseline (single time point during study visit)
  Calculated insulin resistance based on fasting glucose and insulin levels in study participants.
Hormonal Profiles (FSH, LH, AMH, Total and Free Testosterone) | At baseline (single time point during study visit)
  Measurement of key reproductive hormone levels by electrochemiluminescence immunoassay to assess endocrine function in PCOS and control groups.
Ovarian Volume | At baseline (single time point during study visit)
  Ovarian volume measured by standardized transabdominal or transvaginal ultrasonography using the ellipsoid formula.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Gayhan, Medicine, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakıf University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
At this time, a definitive plan for sharing individual participant data (IPD) has not been finalized. The study team acknowledges the importance of data sharing for scientific transparency and collaboration and will evaluate the feasibility and ethical considerations related to IPD sharing following study completion. Any future plans for data sharing will comply with applicable privacy regulations and institutional policies.

REFERENCES:
- [Background] Kara O, Arsoy HA, Keskin M. Relationship between nonalcoholic fatty liver disease and hyperandrogenemia in adolescents with polycystic ovary syndrome. Clin Exp Pediatr. 2023 Sep;66(9):395-402. doi: 10.3345/cep.2023.00353. Epub 2023 Jun 14. PMID 37321582
- [Background] Macut D, Tziomalos K, Bozic-Antic I, Bjekic-Macut J, Katsikis I, Papadakis E, Andric Z, Panidis D. Non-alcoholic fatty liver disease is associated with insulin resistance and lipid accumulation product in women with polycystic ovary syndrome. Hum Reprod. 2016 Jun;31(6):1347-53. doi: 10.1093/humrep/dew076. Epub 2016 Apr 12. PMID 27076501
- [Background] Taranto DOL, Guimaraes TCM, Couto CA, Candido AL, Azevedo RCS, Mattos FS, Elias MLC, Reis FM, Rocha ALL, Faria LC. Nonalcoholic fatty liver disease in women with polycystic ovary syndrome: associated factors and noninvasive fibrosis staging in a single Brazilian center. Arch Endocrinol Metab. 2020 May-Jun;64(3):235-242. doi: 10.20945/2359-3997000000242. PMID 32555989
- [Background] Petta S, Ciresi A, Bianco J, Geraci V, Boemi R, Galvano L, Magliozzo F, Merlino G, Craxi A, Giordano C. Insulin resistance and hyperandrogenism drive steatosis and fibrosis risk in young females with PCOS. PLoS One. 2017 Nov 21;12(11):e0186136. doi: 10.1371/journal.pone.0186136. eCollection 2017. PMID 29161258
- [Background] Chen W, Pang Y. Metabolic Syndrome and PCOS: Pathogenesis and the Role of Metabolites. Metabolites. 2021 Dec 14;11(12):869. doi: 10.3390/metabo11120869. PMID 34940628
- [Background] Migacz M, Pluta D, Baranski K, Krajewski B, Madej P, Holecki M. Using non-invasive indicators to screen the PCOS population for liver disease - a single-centre study. Endokrynol Pol. 2025;76(1):94-99. doi: 10.5603/ep.101901. PMID 40071805
- [Result] Chakraborty S, Ganie MA, Masoodi I, Jana M; Shalimar; Gupta N, Sofi NY. Fibroscan as a non-invasive predictor of hepatic steatosis in women with polycystic ovary syndrome. Indian J Med Res. 2020 Apr;151(4):333-341. doi: 10.4103/ijmr.IJMR_610_18. PMID 32461397
- See also: Study examining the relationship between nonalcoholic fatty liver disease and hyperandrogenemia in adolescents with PCOS. — https://pubmed.ncbi.nlm.nih.gov/37321582/
- See also: Research on the association of NAFLD with insulin resistance and lipid accumulation in women with PCOS. — https://pubmed.ncbi.nlm.nih.gov/27076501/